CLINICAL TRIAL: NCT06585449
Title: A Randomized, Double-blind, Placebo-controlled Study, to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intrathecally Administered Single Ascending Doses of ALN-HTT02 in Adult Patients With Huntington's Disease
Brief Title: A Study to Evaluate ALN-HTT02 in Adult Patients With Huntington's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALN-HTT02-001
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Huntington's Disease
Keywords: siRNA; ALN-HTT02; Intrathecal; HD-ISS Stage 2; HD-ISS early Stage 3; Neurodegenerative disorder
MeSH Terms: conditions — Huntington Disease; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ALN-HTT02 (Experimental): Participants will be administered a single dose of ALN-HTT02 during the Double-blind Part of the study. Participants who received ALN-HTT02 in the Double-blind part of the study will not receive an additional dose during the Open-label part of the study
  Interventions: Drug: ALN-HTT02
- Placebo + ALN-HTT02 (Placebo Comparator): Participants will be administered a single dose of placebo during the Double-blind Part of the study. Participants will have the option to receive a single dose of ALN-HTT02 during the Open-Label Part of the study.
  Interventions: Drug: ALN-HTT02; Drug: Placebo

INTERVENTIONS:
Drug: ALN-HTT02 — ALN-HTT02 will be administered intrathecally
Drug: Placebo — Placebo will be administered intrathecally
  Arms: Placebo + ALN-HTT02

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacodynamics (PD) and pharmacokinetics (PK) of a single dose of ALN-HTT02.

ELIGIBILITY:
Inclusion Criteria

* Has stage 2 or early Stage 3 Huntington's disease (HD), per the Huntington's Disease Integrated Staging System (HD-ISS)

Exclusion Criteria

* Has significant structural or degenerative neurologic disease other than Huntington's Disease (HD) at screening
* Has primary or secondary immune compromise at screening due to infections, medical conditions, or chronic therapies
* Has alanine aminotransferase or aspartate aminotransferase >2× upper limit of normal (ULN)
* Has an estimated glomerular filtration rate (eGFR) of <45 mL/min/1.73m^2 at screening
* Has received an investigational agent within the last 1 year or 5 half-lives (if known)

Note: other protocol defined inclusion / exclusion criteria apply

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2028-07-05 (Estimated); Study Completion 2028-07-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) in the Double-blind Part of the Study | Up to 12 months
Frequency of AEs in the Open-label Part of the Study | Up to 12 months

SECONDARY OUTCOMES:
Change from Baseline in Levels of Mutant Huntingtin (mHTT) in Cerebrospinal Fluid (CSF) | Baseline up to Month 12 in the Double-blind Part of the study; Baseline up to Month 12 in the Open-label Part of the study
Concentrations of ALN-HTT02 in Plasma | Up to Month 12 in the Double-blind Part of the study; Up to Month 12 in the Open-label Part of the study
  Area Under the Plasma Concentration-time Curve (AUC) Maximum Observed Plasma Concentration (Cmax) Time to Maximum Plasma Concentration (Tmax)
Concentrations of ALN-HTT02 in Cerebrospinal Fluid (CSF) | Up to Month 12 in the Double-blind Part of the study; Up to Month 12 in the Open-label Part of the study
Concentrations of ALN-HTT02 in Urine | Up to Month 12 in the Double-blind Part of the study; Up to Month 12 in the Open-label Part of the study
  Fractional Excretion of ALN-HTT02

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (19):
- Canada (4):
  - Clinical Trial Site, Edmonton, Alberta
  - Clinical Trial Site, Vancouver, British Columbia
  - Clinical Trial Site, Ottawa, Ontario
  - Clinical Trial Site, Montreal, Quebec
- Germany (7):
  - Clinical Trial Site, Ulm, Baden-Wurttemberg
  - Clinical Trial Site, Taufkirchen, Bavaria
  - Clinical Trial Site, Bochum, Northwest
  - Clinical Trial Site, Bonn, Northwest
  - Clinical Trial Site, Münster, Northwest
  - Clinical Trial Site, Dresden, Saxony
  - Clinical Trial Site, Berlin, State of Berlin
- United Kingdom (8):
  - Clinical Trial Site, Cambridge, CAM
  - Clinical Trial Site, Plymouth, DEV
  - Clinical Trial Site, Glasgow, GLG
  - Clinical Trial Site, London, LND
  - Clinical Trial Site, Manchester, MAN
  - Clinical Trial Site, Oxford, OXF
  - Clinical Trial Site, Cardiff, VGL
  - Clinical Trial Site, Birmingham, WAR

IPD SHARING:
Plan to Share IPD: No